CLINICAL TRIAL: NCT07373444
Title: Westlake Aging Cohort
Brief Title: Westlake Aging Cohort (WeAC)
Status: Not yet recruiting | Type: Observational
Sponsor: Westlake University (Other)
Collaborators: Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University (Unknown); The Third People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 20251023ZJS001
Record Dates: First submitted 2025-12-24; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Aging; Cognition Improvement; Cognition Disorders; Cognition
Keywords: aging; cognition; gut microbiota; multi-omics; brain
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Westlake Ageing Cohort (WeAC) is a longitudinal cohort study conducted in Hangzhou, Zhejiang Province, China. The investigators aim to enroll 2,800 participants aged 55 years and older for long-term follow-up. The population will include individuals with neurodegenerative diseases or those at the prodromal stage of cognitive impairment, as well as healthy middle-aged and older adults serving as controls. The investigators will collect their sociodemographic, dietary, lifestyle, clinical, and neuroimaging data, as well as biological samples.

DETAILED DESCRIPTION:
The investigators will recruit middle-aged and aged participants, including healthy controls and individuals with neurodegenerative disorders such as mild cognitive impairment (MCI), Alzheimer's disease (AD), Parkinson's disease dementia (PDD), and dementia with Lewy bodies (DLB), etc. The aim of this study is to construct a longitudinal database that includes sociodemographic, lifestyle, clinical, neuroimaging, and multi-omics data. This database will be used to characterize the molecular signatures of neurodegenerative disorders. In addition, the investigators will identify biomarkers associated with neurodegenerative diseases. Furthermore, the investigators aim to uncover the mechanisms underlying the progression of mild cognitive impairment (MCI) and other neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 55 and 90 years (inclusive) at baseline.
2. Availability of a companion capable of providing independent functional assessments and fluent in Chinese.
3. Willingness and ability to regularly complete required surveys and physical examinations as per study protocol.
4. MMSE scores were required to be 24-30 (inclusive) for healthy controls and MCI; and 20-24 (inclusive) for AD and DLB/PDD patients.
5. Healthy controls: CDR = 0, memory box = 0. MCI: CDR = 0.5, memory box ≥ 0.5. AD: CDR = 0.5 or 1. The DLB/PDD meets the core features of diagnosis.
6. Healthy controls exhibit no significant cognitive or functional decline. Patients with MCI have objective cognitive impairment not sufficient for an AD diagnosis. AD patients fulfill the NINCDS-ADRDA criteria. DLB/PDD patients meet their respective international consensus diagnostic criteria. Other neurodegenerative diseases meet the diagnostic criteria.

Exclusion Criteria:

1. Participants with major medical or neuropsychiatric conditions unrelated to the study purposes were excluded. These included, but were not limited to, psychiatric disorders, cancer, infectious diseases, structural brain abnormalities, and epilepsy.
2. Current use of psychoactive medications or any other drugs that may affect the study.
3. Participants with cardiac pacemakers, artificial heart valves, or metallic implants in the eyes, skin, or any other part of the body.
4. Participants with any other diseases that may affect the study.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants must be Chinese residents, regardless of their ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 48 months
  Cognitive function will be evaluated using the Mini-Mental State Examination (MMSE, score range: 0-30, with higher scores indicating better cognitive function) and clinical diagnosis provided by physicians.
Gut microbiome | 48 months
  The gut microbiome will be profiled by metagenomic sequencing or ITS rRNA sequencing. In addition, fecal microbiota will be cultured, isolated, and identified.

SECONDARY OUTCOMES:
Brain magnetic resonance imaging | 48 months
  Use brain magnetic resonance imaging (MRI) to measure the brain structure and function of participants.
Positron emission tomography | 48 months
  Assess the brain function and neurological disorders by positron emission tomography (PET).
Brain images relevant inspections | 48 months
  Other brain image relevant inspections required for study to measure brain structure and function of participants.
Electroencephalogram | 48 months
  Electroencephalogram (EEG) monitors the electrical activity of the brain. And further measure based on coupled EEG/MEG and eye-tracking.
Blood biochemical parameters | 48 months
  Blood biochemical parameters, including glucose and lipids, will be analyzed using an automated biochemical analyzer.
Serum inflammatory factors | 48 months
  Detect and assess serum inflammatory factors such as IL-1β, IL-6, and IL-12, in serum from participants.
Health and behavior monitoring | 48 months
  Use fitness trackers to record the physiological and behavioral data of participants.
Sleep data measurement | 48 months
  Use the polysomnography (PSG) to record the sleep data of participants to evaluate the sleep quality.
Continuous glucose monitoring | 48 months
  Use the continuous glucose monitoring (CGM) for dynamic blood glucose recording to determine the glycemic control of participants.
Environmental measurement | 48 months
  Use the environmental monitoring device to measure various exposure factors in the participants' living environment.
Multi-omics data | 48 months
  Multi omics results of detecting biological samples such as plasma, peripheral blood mononuclear cells (PBMCs), urine, feces, saliva, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (2):
- China (2):
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided